CLINICAL TRIAL: NCT07344428
Title: Therapeutic Effect of Exclusion Diet Combined With Anti-TNF-α Biologics in Adult Patients With Crohn's Disease in China: A Single-center, Prospective, Randomized, Controlled Trial
Brief Title: Efficacy and Safety of CDED With Anti-TNF-α Biologics in Crohn's Disease: A Randomized Trial
Acronym: CDED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021ZSLYEC-127-CDED
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Crohn's Disease；Mucosal Healing；Dietary Intervention
Keywords: Crohn's Disease, exclusion diet, biologics, randomized controlled trial
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crohn's Disease Exclusion Diet + Anti-TNF-α biologics (Experimental): Participants in this group will receive anti-TNF-α biologics (infliximab 5mg/kg IV at weeks 0, 2, 6, and 14, or adalimumab subcutaneous injection at standard doses) combined with the Crohn's Disease Exclusion Diet (CDED). The CDED protocol includes detailed dietary guidance specifying allowed foods (rice, certain vegetables and fruits, fish, poultry, olive oil) and prohibited items (ultra-processed foods, nuts, legumes, butter). Patients will maintain daily food diaries and receive frequent supervision and guidance from researchers to ensure dietary compliance.
  Interventions: Other: Crohn's Disease Exclusion Diet
- Anti-TNF-α biologics only (No Intervention): Participants in this group will receive anti-TNF-α biologics alone (infliximab 5mg/kg IV at weeks 0, 2, 6, and 14, or adalimumab subcutaneous injection at standard doses) without any dietary intervention. This group serves as the control to evaluate the additional benefit of CDED when combined with standard biologic therapy. No specific dietary restrictions or guidance will be provided to this group.

INTERVENTIONS:
Other: Crohn's Disease Exclusion Diet — Participants will receive anti-TNF-α biologics (infliximab 5mg/kg IV at weeks 0, 2, 6, and 14, or adalimumab subcutaneous injection at standard doses) combined with the Crohn's Disease Exclusion Diet (CDED). The CDED protocol includes detailed dietary guidance specifying allowed foods (rice, certain vegetables and fruits, fish, poultry, olive oil) and prohibited items (ultra-processed foods, nuts, legumes, butter). Patients will maintain daily food diaries and receive frequent supervision and guidance from researchers to ensure dietary compliance throughout the 14-week study period. This combined intervention aims to evaluate whether CDED can synergistically enhance the efficacy of standard biologic therapy in achieving mucosal healing in Crohn's disease patients.
  Arms: Crohn's Disease Exclusion Diet + Anti-TNF-α biologics

SUMMARY:
Crohn's disease (CD) is a chronic inflammatory bowel disease with high recurrence and surgical rates. Mucosal healing is a key therapeutic goal, yet current anti-TNF-α biologics achieve only about 30% mucosal healing. Dietary intervention, particularly the Crohn's Disease Exclusion Diet (CDED), shows promise in CD management. Preliminary data suggest that combining CDED with anti-TNF-α biologics may significantly improve mucosal healing rates (42.9% vs 25%). This single-center, prospective, randomized, controlled trial will enroll 185 adult CD patients with active disease (SES-CD ≥3), randomly assigned 1:1 to receive either anti-TNF-α biologics plus CDED or anti-TNF-α biologics alone. The primary endpoint is mucosal healing rate at week 14 (SES-CD=0). Secondary endpoints include clinical remission, endoscopic response, transmural healing, and adverse events. This study aims to provide high-quality evidence for the efficacy and safety of this combined approach in Chinese CD patients.

DETAILED DESCRIPTION:
Crohn's disease (CD) is a chronic granulomatous inflammatory disease that can affect the entire digestive tract, characterized by a protracted course and complex complications. Although the advent of biologics has significantly improved CD treatment outcomes, real-world data show that only about 30% of patients achieve mucosal healing with anti-TNF-α biologics (infliximab or adalimumab), representing a major therapeutic bottleneck. According to the international STRIDE-II consensus, mucosal healing is a key target in CD treat-to-target strategy and is closely associated with better long-term prognosis. In recent years, the role of dietary factors in CD management has gained increasing attention. Exclusive enteral nutrition (EEN) has demonstrated efficacy in inducing remission and mucosal healing in pediatric CD, but poor long-term adherence limits its application in adults. Based on this, oral dietary regimens mimicking EEN components (such as the Crohn's Disease Exclusion Diet, CDED) have become a new research focus. Preliminary data from our research team showed that compared to anti-TNF-α biologics alone, CDED combined with anti-TNF-α biologics resulted in significantly higher mucosal healing rates (42.9% vs 25.0%) and greater improvement in SES-CD scores at week 14, providing strong preliminary evidence for this combined approach to overcome the efficacy bottleneck.This is a single-center, prospective, randomized, open-label, controlled clinical trial conducted at the Inflammatory Bowel Disease Center, Department of Gastroenterology, Sixth Affiliated Hospital of Sun Yat-sen University. A total of 185 eligible adult Chinese patients with active CD will be enrolled and randomly assigned in a 1:1 ratio using SAS-generated random sequences with sealed envelope allocation concealment. The intervention group will receive standardized anti-TNF-α biologic therapy (infliximab 5mg/kg IV at weeks 0, 2, 6, and 14, or adalimumab subcutaneous injection at standard doses) combined with strict CDED. The dietary protocol includes detailed electronic and paper recipes specifying allowed grains (rice only), vegetables (avoiding nightshades), fruits, meats (recommended fish and poultry, limited red meat), oils (olive oil, coconut oil), and cooking methods (steaming, boiling, blanching), while strictly prohibiting ultra-processed foods, nuts, legumes, and butter. Patients will maintain daily food diaries via WeChat group and shared documents, with frequent supervision and guidance from researchers. The control group will receive the same anti-TNF-α biologic therapy alone without dietary intervention. The primary endpoint is mucosal healing rate at week 14 (defined as SES-CD score=0). Secondary endpoints include clinical remission rate (CDAI<150), endoscopic response rate (≥50% reduction in SES-CD), transmural healing rate (assessed by intestinal ultrasound), and adverse event incidence. Sample size calculation is based on preliminary data with superiority test assumption and 20% dropout rate. Data analysis will follow intention-to-treat (ITT) principle using SPSS 25.0 software.This study is innovative as it is the first in China to use a rigorous randomized controlled trial design to validate whether a specific, easily implementable, and cost-effective dietary intervention (CDED) can synergistically enhance the efficacy of standard biologic therapy, aiming to overcome the limitation of suboptimal mucosal healing rates with biologics alone. The findings are expected to provide high-level evidence for long-term dietary management in CD patients, forming a dietary intervention guidance program with Chinese characteristics, thereby improving patient outcomes and reducing healthcare burden.

ELIGIBILITY:
Inclusion Criteria:1.Age: Aged ≥18 years.2.Diagnosis: Diagnosis of Crohn's disease confirmed by endoscopy and histopathology, with active disease (CDAI ≥150).3.Treatment Indication: Indicated for anti-TNF-α biologic therapy (infliximab or adalimumab) and being naive to these specific agents.4.Informed Consent: Willing and able to provide written informed consent.5.Compliance: Able to understand and comply with the study protocol requirements, including dietary intervention and follow-up schedule.

-

Exclusion Criteria:1.Severe Complications: Presence of intestinal obstruction, intra-abdominal abscess, intestinal fistula, or other severe complications requiring surgical intervention.2.Comorbidities: Severe cardiac, hepatic, or renal insufficiency (e.g., Child-Pugh class C, or eGFR <30 mL/min/1.73 m²).3.Infection Risk: Active tuberculosis, active hepatitis B, HIV infection, or other severe opportunistic infections.4.Malignancy: Current or history of malignancy, except for non-melanoma skin cancer.5.Pregnancy Status: Pregnant or breastfeeding women, or women planning pregnancy during the study period.6.Medication Use: Recent use (within 3 months) of other immunosuppressants (e.g., azathioprine, methotrexate) or corticosteroids (e.g., prednisone >20 mg/day).7.Dietary Restrictions: Severe food allergies, celiac disease, severe malnutrition (BMI <18.5 kg/m²), or inability to adhere to the Crohn's Disease Exclusion Diet (CDED).8.Other Factors: Concurrent participation in another clinical trial, or any other condition deemed by the investigator to make the patient unsuitable for study participation.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Mucosal healing rate at week 14 (SES-CD=0) | Week 14 (from baseline to week 14)
  The proportion of patients achieving complete mucosal healing, defined as a Simple Endoscopic Score for Crohn's Disease (SES-CD) score of 0 at week 14. SES-CD is a validated endoscopic scoring system that assesses the severity of mucosal inflammation in Crohn's disease, evaluating four parameters: ulcer size, ulcerated surface, affected surface, and presence of stenosis. A score of 0 indicates no visible inflammation or ulceration in the entire colon and terminal ileum, representing complete mucosal healing. Endoscopic assessments will be performed by experienced gastroenterologists who are blinded to treatment allocation.

SECONDARY OUTCOMES:
Clinical remission rate at week 14 (CDAI<150) | Week 14 (from baseline to week 14)
  The proportion of patients achieving clinical remission, defined as a Crohn's Disease Activity Index (CDAI) score less than 150 at week 14. CDAI is a validated clinical scoring system that evaluates eight parameters including number of liquid stools, abdominal pain, general well-being, extraintestinal manifestations, use of antidiarrheals, abdominal mass, hematocrit, and body weight. A score below 150 indicates clinical remission. Assessments will be performed by trained clinicians at each study visit.
Endoscopic response rate at week 14 (SES-CD reduction ≥50%) | Week 14 (from baseline to week 14)
  The proportion of patients achieving endoscopic response, defined as a reduction of at least 50% in the Simple Endoscopic Score for Crohn's Disease (SES-CD) from baseline to week 14. SES-CD evaluates four endoscopic parameters in five colonic segments: ulcer size, ulcerated surface, affected surface, and presence of stenosis. A 50% reduction in total score indicates significant improvement in mucosal inflammation. Endoscopic evaluations will be conducted by blinded gastroenterologists.
Transmural healing rate at week 14 (intestinal ultrasound) | Week 14 (from baseline to week 14)
  The proportion of patients achieving transmural healing, assessed by intestinal ultrasound with a maximum bowel wall thickness ≤3mm and absence of inflammatory signs. Transmural healing is defined as the normalization of bowel wall thickness and the resolution of inflammatory changes in the entire intestinal wall layers. Ultrasound examinations will be performed by experienced radiologists blinded to treatment allocation using standardized protocols.
Incidence of adverse events during 14-week treatment period | Week 14 (from baseline to week 14)
  The incidence of all adverse events including diet-related malnutrition, allergic reactions, infusion reactions, injection site reactions, opportunistic infections, and other treatment-emergent adverse events. Adverse events will be monitored throughout the study period and graded according to the National Institute on Aging (NIA) severity criteria. Causality assessment will be performed by investigators using standardized criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Sixth afflicated of Sun-yat sen university, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No